CLINICAL TRIAL: NCT02268539
Title: Efficacy, Safety and Efficiency of the nMARQ Pulmonary Vein Isolation System in the Treatment of Paroxysmal Atrial Fibrillation - A Pilot Study
Brief Title: Efficacy, Safety and Efficiency of the nMARQ Pulmonary Vein Isolation System in Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: B703
Record Dates: First submitted 2014-07-22; First posted 2014-10-20 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: pilot study; atrial fibrillation; ablation; implanted loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ablation at 20 watt / 30 seconds (Active Comparator): Participants randomised to 20 watt ablation for 30 seconds
  Interventions: Procedure: ablation
- Ablation at 20 watt /45 seconds (Active Comparator): 20 watt ablation for 45 seconds
  Interventions: Procedure: ablation
- Ablation at 25 watt / 30 seconds (Active Comparator): 25 watt ablation for 30 seconds
  Interventions: Procedure: ablation
- iAblation at 25 watt / 45 seconds (Active Comparator): 25 watt ablation for 45 seconds
  Interventions: Procedure: ablation

INTERVENTIONS:
Procedure: ablation — Ablation ranging from 20-25 watts / 30-45 seconds

SUMMARY:
This is a pilot study designed to investigate the effectiveness of the nMARQ Pulmonary Vein Isolation system in the treatment of Paroxysmal Atrial Fibrillation (AF) at different ablation settings.

AF is a common condition which causes a fast and erratic heartbeat. There are estimated to be 50,000 new cases diagnosed per year in the UK. The fast heart beat can cause symptoms such as palpitations, lightheadedness, chest pains, shortness of breath and fatigue.

Catheter ablation is a technique used for the control of AF. In this procedure a catheter (a long thin wire) is passed into the chambers of the heart via a large blood vessel in a leg. The tip of the catheter can destroy tiny sections of heart tissue that may be the source or trigger of the abnormal electrical impulses. One of the challenges of AF ablation is to maximize success rates, as such there is currently rapid advances in technology to carry out this procedure.

Different catheters exist which deliver this energy in different ways. This study uses one such system to perform this procedure. It is called the nMARQ system for Pulmonary Vein Isolation produced by Biosense Webster. Currently this system is used in practice in the UK for patients with this medical condition.

What we seek to research is when ablating what is the optimum setting to perform ablation at. There is currently no data to guide best clinical practice in this area.

DETAILED DESCRIPTION:
This is a pilot study designed to investigate the use of the nMARQ Pulmonary Vein Isolation system in the treatment of Paroxysmal Atrial Fibrillation (AF) at different ablation settings.

At least one month prior to the ablation procedure, an Implanted Loop Recorder (ILR) (the REVEAL XT) will be implanted into the patient for robust, continuous, long term monitoring of the burden of arrhythmia following the case.

It has been decided to use continuous implanted rhythm monitors to allow for robust complete data capture of arrhythmia recurrence and burden with little impact to the patient after implantation. These are increasingly being used in the follow up of patients undergoing AF ablation. They give a continuous data feed showing the presence and quantity of abnormal rhythm seen after ablation. Their use has been approved in the follow up of AF ablation procedures within recent consensus guidelines formulated by the American College of Cardiology, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, and the Heart Rhythm Society. There are several papers showing the validation of data collected by the REVEAL XT ILR and the benefit of continuous monitoring versus conventional methods of intermittent ambulatory ECGs.

The settings chosen for ablation are guided both by preclinical data collected by Biosense Webster and also the settings being used clinically worldwide when utilising this system. It has been decided to have a two by two study design varying the wattages 20W and 25W and also varying the time periods per lesion 20 seconds and 40 seconds.

We feel that this project can be carried out as a pilot study to potentially inform further research. There is very little clinical data published on how best to use of this device. At present it is left to individual clinicians to form their own "best practise" when choosing ablation settings. We seek to formalise the potential ablation variables into a structured format that will allow for comparisons to be drawn at the end of the study and to form the basis of future research.

Following the current pathway, patients are admitted 24 hours prior to their treatment for further, standard, tests (including an Echo TOE and pregnancy test); at this point patients will be randomised to one of the arms of the trial, at an equal 1:1:1:1 ratio. As the study is ' unblinded ' and the procedure constitute standard care in the NHS , it would be at this point that the participant and Consultant have time to discuss the impact of the setting that the participant has been randomised to, thereby reducing any anxiety on the day of the procedure.

The following day, the procedure would be carried according to standard treatment and following national guidelines using one of the ablation presets as per randomisation.

Within the UK it is standard practice to have a follow-up visit at 6 weeks, 3 months, 6 months and 12 months. At each visit, in addition to the standard tests, the patient and Consultant would complete questionnaires.

After one year the patient will attend for removal of the ILR unless it is deemed to have clinical use for them.

Recruitment and Consent Our target population will be patients who would routinely be having catheter ablation of their AF. They will have the kind of AF that comes and goes and will be troubled symptomatically by it. This research study has been constructed around a patients' normal care pathway, minimising the need for additional visits or activities.

Risks, burdens and benefits Potential risks and burden of participation in the study centre on the use of the ILR for rhythm recording both before and after the ablation procedure. This device is small and implantation is a minor day case procedure done under local anaesthetic. The risk of implantation is very small. Its use in the follow up after AF ablation is endorsed by international clinical guidelines and backed up by scientific data. The use of the ILR after AF ablation is becoming more commonplace and if anything is constrained by financial issues in the NHS rather than any ethical considerations about the risks or burdens of implantation.

Potential benefit to the participant also involves the ILR. By having a continuous monitor of heart rhythm after ablation the consultant has information that can guide clinical management decision making after the ablation occurs. In clinical practise, without the ILR in place, the patient would otherwise have to undergo a number of ambulatory ECG monitors periodically throughout the follow up period

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Symptomatic Paroxysmal Atrial Fibrillation
* Drug refractory to one or more antiarrhythmic medication
* 1st Procedure for Patients
* LA <5.5cm (TTE)

Exclusion Criteria:

* LV EF <30%
* Patient with correctable cause of AF
* Previous cardiac surgery
* History of previous CVA
* Pregnancy
* Smoke or LAA thrombus seen in LA on pre-procedural TOE
* Sub-therapeutic warfarinisation
* Contraindication to formal anticoagulation
* Life expectancy less than 365 days (12 months).
* Enrolment in an investigational study evaluating another device or drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy; freedom from AF at 12 months | One year success
  One year success is defined as freedom from AF/AFL/AT off antiarrhythmic drug therapy as assessed from the end of the 3-month blanking period to 12 months following the ablation procedure in the intention to treat (ITT) population as randomized (based on ILR data)

SECONDARY OUTCOMES:
Safety | 7 days
  Incidence of early-onset primary adverse events within 7 days of the atrial fibrillation ablation procedure and any diagnosed during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Tan, MB BC, MRCP, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No